CLINICAL TRIAL: NCT05165290
Title: Prospective, Double-masked, Randomized, Multi-center, Active-controlled, Parallel-group, 3-month Study Assessing the Safety & Ocular Hypotensive Efficacy of TC-002 Ophthalmic Solution Compared to Latanoprost Ophthalmic Solution 0.005% in Subjects With Elevated Intraocular Pressure
Acronym: TC-002-301
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TearClear Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TC-002-301
Record Dates: First submitted 2021-12-17; First posted 2021-12-21 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Elevated Intraocular Pressure
Keywords: elevated IOP; open-angle glaucoma; ocular hypertension
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment assignments will be masked to the Sponsor, subjects, Investigators and select investigative staff, until completion of the study and the final database is locked. The appearance of the bottles in the two treatment arms are not identical; however, the cartons and labeling on the cartons in which the bottles are supplied will be identical and identified with unique kit numbers. Therefore, the dedicated dosing coordinator will handle IP-related responsibilities but will be otherwise uninvolved in study assessments.
  Appropriate precautions must be taken to prevent unauthorized access to the randomization scheme. Unless the subject's safety requires otherwise and if time permits, the decision to unmask an individual subject's treatment assignment is to be made jointly by the Investigator and Sponsor's medical monitor after consultation with the Sponsor, thus leaving the masking of the remaining subjects intact.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LAT, 0.005% (Active Comparator): Commercially available FDA-approved generic latanoprost ophthalmic solution, 0.005%
  Interventions: Drug: Latanoprost ophthalmic solution, 0.005%
- TC-002 (Experimental): TC-002, TearClear latanoprost ophthalmic solution, 0.005%
  Interventions: Drug: TC-002 latanoprost ophthalmic solution, 0.005%

INTERVENTIONS:
Drug: Latanoprost ophthalmic solution, 0.005% — Commercially available, FDA-approved generic latanoprost ophthalmic solution, 0.005% (LAT) without modification will be used as the active control
  Arms: LAT, 0.005%
Drug: TC-002 latanoprost ophthalmic solution, 0.005% — TC-002 is formulated using the commercially available latanoprost drug substance; delivered drop to the eye is preservative-free.
  Arms: TC-002

SUMMARY:
Prospective, double-masked, randomized, multi-center, active-controlled, parallel-group, 3-month study assessing the safety and ocular hypotensive efficacy of TearClear latanoprost Ophthalmic Solution, 0.005% (TC-002) compared to latanoprost Ophthalmic Solution, 0.005% (LAT) in subjects with elevated intraocular pressure at approximately 20 study sites located in the United States

DETAILED DESCRIPTION:
This is a Phase 3, randomized, investigator-masked, multicenter, parallel-group trial comparing two ophthalmic solution formulations of latanoprost at a fixed dose of 0.005% administered once daily (QD) for 12 weeks.

Approximately 300 subjects will be randomized in this study at approximately 20 sites in the United States (US).

Treatment assignments will be masked to TearClear, study subjects, Investigators and site staff. Because the container closure for the investigational product is different, this study will use an unmasked dosing coordinator at each study site. All clinical trial supplies will be masked by using carton boxes to mask the appearance of the immediate container closure.

At approximately 2 select sites, approximately10% of total randomized subjects will have systemic PK labs drawn.

The study involves 7 clinic visits, including Screening (Visit 1), Randomization (Visit 2) and treatment visits (Visits 3, 5 and 7, during which ophthalmic assessments will occur and IOP will be assessed diurnally. There will be two interim IP dispensation visits (Visits 4 and 6).

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years old.
2. Have been diagnosed and treated for bilateral open-angle glaucoma or ocular hypertension in both eyes.
3. Currently and for at least 30 days prior to screening, are being treated with a stable dose of latanoprost ophthalmic solution or prostaglandin analog for which there is a documented and positive treatment response with either agent maintained within both eyes.
4. Have best corrected visual acuity (BCVA) via Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) score +0.6 logarithm of the minimum angle of resolution (logMAR) or better in each eye.
5. At Visit 1, have IOP on prostaglandin or prostaglandin analog single therapy ≤ 21mmHg, at Visit 2, have diurnal IOP between 22 and 30 mmHG, inclusive for each eye.
6. In the Investigator's judgment, are able to safely discontinue current ocular hypotensive medication during the washout period.
7. Willing and able to avoid wearing contact lenses from Visit 1 (Screening) and for the duration of the trial.
8. Willing and able to self-administer or have an able person available on a daily basis to assist with administration of study medication.
9. Female subjects must either be incapable of pregnancy because of bilateral oophorectomy, hysterectomy, or bilateral tubal ligation, or be post-menopausal (have been amenorrheic for at least 2 years) or must use an effective (e.g., double-barrier) method of birth control for the duration of the study. Female subjects of childbearing potential must have a negative pregnancy test and not be nursing.
10. Willing and able to comply with all study procedures.

Exclusion Criteria:

1. Causes of glaucoma other than primary open-angle glaucoma, including:

   1. narrow angles (3 quadrants with less than Grade 2 according to Shaffer anterior chamber angle grading system) and subjects with angle closure
   2. clinically significant peripheral anterior synechiae
   3. congenital glaucoma
   4. a history of angle closure in either eye
   5. aphakic glaucoma
   6. traumatic glaucoma
   7. neovascular glaucoma
   8. pigmentary glaucoma
   9. pseudoexfoliative glaucoma
   10. drug-induced glaucoma
2. Using a multi-drop treatment (other than prostaglandin or prostaglandin analog) for IOP-lowering medications.
3. Advanced glaucoma or subjects with a cup/disc ratio greater than 0.8.
4. Have undergone incisional IOP-lowering surgeries a placement or removal of minimally invasive glaucoma implant (MIG) in either eye.
5. Have undergone non-incisional IOP-lowering surgeries within the past 6 months.
6. Used anti-vascular endothelial growth factor (anti-VEGF) within 12 months of screening.
7. Used intraocular, periocular or topical corticosteroids within 60 days of screening.
8. Have received laser surgery for glaucoma (selective laser trabeculoplasty [SLT] or argon laser trabeculoplasty [ALT]) within 6 months of screening.
9. Have uveitis, iritis or congenital aphakia.
10. Are unwilling to discontinue current glaucoma medication within 30 days of the randomization (Visit 2).
11. Have had intraocular or periocular surgery within the past 3 months.
12. Are non-responsive to topical prostaglandins, prostamides or prostaglandin analogs in the Investigator's judgement.
13. History of previous complicated cataract surgery, or previous refractive keratotomy in either eye.
14. Used miotics and oral/topical carbonic anhydrase inhibitors within 5 days of screening.
15. Have any known hypersensitivity to any components of the formulation or latanoprost.
16. Have participated in a clinical trial for IOP-lowering investigational product or exposure to an IP within the prior 30 days.
17. In the judgement of the Investigator, have previous or currently active clinically significant systemic or ocular disease in either eye that could affect study outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint is the difference in mean change from baseline (CFB) in IOP | Weeks 2, 6, and 12 at 8:00 AM, 10:00 AM, and 4:00 PM.

SECONDARY OUTCOMES:
Secondary efficacy endpoints include diurnal (average of 8:00 AM, 10:00 AM, and 4:00 PM measurements) IOP | Weeks 2, 6, and 12.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - Global Research Management, Glendale, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Michael K. Tran, MD, Westminster, California
  - Segal Drug Trials, Delray Beach, Florida
  - Shettle Eye Research Inc., Largo, Florida
  - International Research Center, Tampa, Florida
  - The Eyecare Institute/Butcherton Clinical Trials, Louisville, Kentucky
  - Rochester Ophthalmological Group PA, Rochester, New York
  - Abrams Eye Center, Cleveland, Ohio
  - Scott & Christie Associates PC, Cranberry Township, Pennsylvania
  - Total Eye Care P.A., Memphis, Tennessee
  - Louis M. Alpern, M.D., M.P.H., P.A., El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - R&R Research LLC, San Antonio, Texas
  - San Antonio Eye Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No